CLINICAL TRIAL: NCT05118737
Title: Adding Colchicine to Tocilizumab in Hospitalized Patients With Severe COVID-19 Pneumonia: An Open-Label Randomized Controlled Trial
Brief Title: Adding Colchicine to Tocilizumab in Patients With Severe COVID-19 Pneumonia.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRC-01-21-299
Record Dates: First submitted 2021-11-11; First posted 2021-11-12 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-10

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19 Pneumonia; Cholchicin
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: - To evaluate the efficacy of colchicine versus no colchicine in terms of the need of invasive mechanical ventilation among patients with severe COVID-19 pneumonia who received tocilizumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- colchicine (Active Comparator): Intervention arm: colchicine to be used among COVID-19 patients admitted to HMGH, CH, and CDC and already received tocilizumab
  Interventions: Drug: Colchicine
- Control (Placebo Comparator): COVID-19 patients admitted to HMGH, CH, and CDC and already received tocilizumab according to local protocol
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — colchicine to be used among COVID-19 patients admitted to HMGH, CH, and CDC and already received tocilizumab
  Other Names: Colcrys

SUMMARY:
Colchicine acts upstream in the cytokines cascade by inhibiting the NLRP3 inflammasome while IL-6 receptor antagonists (tocilizumab) block the end result of the cytokines cascade. Hence, adding colchicine to tocilizumab with the aim of blocking the early and end products of the cytokines cascade, might reduce the risk of developing cytokine storm and hence the need for invasive mechanical ventilation and eventually death. Therefore, investigators aim to conduct an open-label randomized controlled trial to evaluate the efficacy and safety of adding colchicine to tocilizumab among patients with severe COVID-19 pneumonia in an attempt to reduce the rate of invasive mechanical ventilation and mortality. Investigators will include patients with severe COVID-19 pneumonia and already received tocilizumab according to local protocol. Enrolled patient will be then randomized in 1:1 to colchicine versus no colchicine. Patients will be followed up until discharge or for 30 days, whichever comes first. Data will be collected from electronic medical profiles. The primary efficacy outcome will be rate of invasive mechanical ventilation and will be determined using Cox proportional hazard model.

DETAILED DESCRIPTION:
The novel coronavirus infection (COVID-19) significantly contributes to increased mortality in many countries, with a continuously increasing number of infected cases worldwide.1 As of the end of February 2021, there have been over 112 million confirmed cases of COVID-19, including 2.5 million deaths globally.2 The leading cause of mortality due to COVID-19 is respiratory failure from acute respiratory distress syndrome (ARDS).3 The mechanisms by which COVID-19 induces ARDS is currently thought to be due to the activation of the innate immune system leading to hypercytokinemia and hence cytokine storm.

COVID-19 disease course can be divided into three phases; (1) early infection phase, where the virus penetrates host cells in the lung parenchyma; (2) pulmonary phase, in which the viral propagation causes lung tissue injury and hence the host immune response is activated; and (3) the inflammatory cascade, which is triggered by the viral RNA and it is comprised of inflammasome activation that drives the cytokine storm.4,5 SARS-CoV-2 acts on the macrophages to release the nod-like receptor protein 3 (NLRP3) inflammasome, leading to the conversion of pro-interleukin (IL)-1 and pro-IL-18 to their active forms.6,7 The production of IL-1 leads to IL-6 synthesis which is a cytokine that induces C reactive protein (CRP) and has been considered a major proinflammatory agent in the COVID-19 cytokine storm.8-11 Consequently, a few biological therapies that have been studied and used for the treatment of COVID-19 to target specific cytokines augmented by the disease, including anakinra for IL-1, and tocilizumab for IL-6.

Early in the COVID-19 pandemic, the therapeutic efficacy of IL-6 antagonists was evaluated. So far, the results of the evidence assessing the use of IL-6 antagonists are somewhat controversial. A meta-analysis of seven retrospective observational studies using tocilizumab in patients with severe COVID-19 found that tocilizumab resulted in lower all-cause mortality compared to placebo without achieving statistical significance. Furthermore, the risk of ICU admission and the need for mechanical ventilation were similar between the two groups. Recently, the REMAP-CAP trial evaluated the use of a single injection of an IL-6 receptor blocker, tocilizumab or sarilumab, compared to placebo among 800 patients in need of respiratory or blood-pressure support or both. It showed that IL-6 antagonist resulted in an in-hospital mortality of 27%, as compared with 36% in the control group. On the contrary, the COVACTA trial evaluated the use of tocilizumab versus placebo among 452 patients with severe COVID-19 pneumonia and it showed that the mortality rate was 19.7% in the tocilizumab group versus 19.4% in the control group. Therefore, in the absence of potent antiviral therapies to block SARS-CoV-2 replication, it remains unclear whether blocking IL-6 alone is effective.

Colchicine is one of the oldest anti-inflammatory therapies that is approved for treating and preventing acute gout attacks and familial Mediterranean fever. Colchicine has been shown to interfere with the activation of the NLRP3 inflammasome, reducing IL-1 production, which in turn prevents IL-6 release and neutrophils and macrophages activation. Consequently, colchicine targets multiple cytokines in the inflammatory cascade of the cytokine storm induced by COVID-19, which makes it a potential anti-inflammatory therapy for COVID-19. Colchicine differs from IL-6 receptor blockers by having pleotropic mechanisms of action, acting upstream of the cascade of cytokines, and being an oral agent. A few studies have evaluated the use of colchicine in hospitalized patients with COVID-19. The GRECO-19 trial was the first open-label randomized trial that evaluated the efficacy of colchicine versus usual care in non-critically ill hospitalized patients. The study included 105 patients and found a significant reduction in the primary outcome of a two-point deterioration on World Health Organization disease severity scale. Additionally, in a single center cohort study in Italy, the use of colchicine in 122 hospitalized patients with COVID-19 compared with 140 patients who received hydroxychloroquine and/or intravenous dexamethasone; and/or lopinavir/ritonavir, resulted in a significantly better survival rate at 21 days (84.2% versus 63.6% respectively, p=0.001).22 Moreover, there are a few ongoing trials in different countries evaluating the use of colchicine in COVID-19 in comparison to standard care, while excluding the concurrent use of IL-6 antagonists: Given its ease of use, low cost, good safety profile, having different anti-inflammatory mechanism of action than other IL-6 blockade, and the lack of an effective therapy for COVID-19 so far, colchicine might serve as a potential anti-inflammatory agent among patients with severe COVID-19 pneumonia. Colchicine acts upstream in the cytokines cascade by inhibiting the NLRP3 inflammasome while IL-6 receptor antagonists block the end result of the cytokines cascade. The latter might be the reason behind the controversies surrounding tocilizumab efficacy in treating COVID-19 as it has been thought that the ongoing replication of the virus overwhelms the drug capacity to control the disease burden. Given the lack of potent anti-viral agents against SARS-CoV-2, adding colchicine to tocilizumab with the aim of blocking the early and end products of the cytokines cascade, might reduce the risk of developing cytokine storm and hence the need for invasive mechanical ventilation and eventually death. Therefore, investigators aim to conduct an open-label randomized controlled trial to evaluate the efficacy and safety of adding colchicine to tocilizumab among patients with severe COVID-19 pneumonia in an attempt to reduce the rate of invasive mechanical ventilation and mortality.

ELIGIBILITY:
Inclusion Criteria:

* - Alert and conscious adults with the age of > 18 years old Severe COVID-19 pneumonia

  o SpO2 <94% on room air at sea level, respiratory frequency >30 breaths/min, or lung infiltrates >50%
* Received tocilizumab within 10 days prior to enrollment
* Tocilizumab is co-admisnitered with a systemic corticosteroid
* Agree to sign conflict of interest

Exclusion Criteria:

* - Severe COVID-19 pneumonia requiring invasive mechanical ventilation
* Creatinine clearance < 30 mL/min
* End stage renal disease on hemodialysis
* ALT and/or AST > 5 upper limit of normal
* Pregnancy
* Lactation
* To prevent colchicine toxicity, patients receiving a strong CYP3A4 inhibitor (eg clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, atazanavir), a moderate CYP3A4 inhibitor (eg diltiazem, verapamil, fluconazole, amprenavir, aprepitant, fosamprenavir) or a P-gp Inhibitor (eg cyclosporine, ranolazine), will be excluded

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Rate of invasive mechanical ventilation | 6 months
  Rate of invasive mechanical ventilation among patients who received colchicine versus those who did not receive colchicine

SECONDARY OUTCOMES:
Time to invasive mechanical ventilation | 6 months
  Length of time from admission to mechanical ventilation
Duration of invasive mechanical ventilation | 6 months
  Length of time from intubation to extubation
Mortality | 6 months
  30-day in-hospital mortality
ICU length of stay | 6 months
  ICU length of stay from ICU admission to ICU discharge
Hospital length of stay | 6 months
  Hospital length of stay from hospital admission to hospital discharge
Change in inflammatory markers (CRP) | 6 months
  μg/mL
Change in inflammatory markers, (D-Dimer) | 6 months
  mcg/mL
Change in inflammatory markers( IL-6) | 6 months
  pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Rahhal, Msc, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Alaa Rahal, Doha, DA, Qatar

IPD SHARING:
Plan to Share IPD: No
Not allowed as per organization rules for researches with informed consents